CLINICAL TRIAL: NCT03969758
Title: Efficacy of Empirical Ciprofloxacin Plus Metronidazole and Cefixime Plus Metronidazole Therapy for the Treatment of Liver Abscess: A Randomised Controlled Clinical Trial
Brief Title: Ciprofloxacin Plus Metronidazole Vs Cefixime Plus Metronidazole Therapy for the Treatment of Liver Abscess
Acronym: CMETRO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Deba Prasad Dhibar, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INT/IEC/2019/001028
Record Dates: First submitted 2019-05-22; First posted 2019-05-31 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Liver Abscess
MeSH Terms: conditions — Liver Abscess | interventions — Ciprofloxacin; Metronidazole; Cefixime

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciprofloxacin plus Metronidazole therapy (Active Comparator): Will receive tablet Ciprofloxacin (500 mg BDS) and tablet Metronidazole (800 mg TDS) orally for 2 weeks. Percutaneous aspiration or drainage of the liver abscess will be done for all the participants when there is enough liquid content/pus which is amenable for aspiration or drainage. Percutaneous drainage or aspiration will be done in liver abscess with size of ≥ 5 cm and <5 cm respectively. After 2 weeks of empirical antibiotic therapy, asymptomatic patients with persistent drainage with USG showing significant drainable collection in the liver will receive another 2 weeks of extended antimicrobial therapy of same combination.
  Interventions: Drug: Ciprofloxacin
- Cefixime plus Metronidazole Therapy (Active Comparator): Will receive tablet Cefixime (200 mg BDS) and tablet Metronidazole (800 mg TDS) orally for 2 weeks.Percutaneous aspiration or drainage of the liver abscess will be done for all the participants when there is enough liquid content/pus which is amenable for aspiration or drainage. Percutaneous drainage or aspiration will be done in liver abscess with size of ≥ 5 cm and <5 cm respectively. After 2 weeks of empirical antibiotic therapy, asymptomatic patients with persistent drainage with USG showing significant drainable collection in the liver will receive another 2 weeks of extended antimicrobial therapy of same combination.
  Interventions: Drug: Cefixime

INTERVENTIONS:
Drug: Ciprofloxacin — will receive tablet Ciprofloxacin (500 mg BDS) and tablet Metronidazole (800 mg TDS) for 2 weeks orally. Percutaneous aspiration or drainage of the liver abscess will be done when there is enough liquid content/pus amenable for aspiration or drainage. Percutaneous drainage or aspiration will be done in liver abscess with size of ≥ 5 cm and <5 cm respectively.
  Other Names: Metronidazole; Percutaneous drainage or aspiration of the liver abscess
  Arms: Ciprofloxacin plus Metronidazole therapy
Drug: Cefixime — will receive tablet Cefixime (200 mg BDS) and tablet Metronidazole (800 mg TDS) for 2 weeks orally. Percutaneous aspiration or drainage of the liver abscess will be done when there is enough liquid content/pus amenable for aspiration or drainage. Percutaneous drainage or aspiration will be done in liver abscess with size of ≥ 5 cm and <5 cm respectively.
  Other Names: Metronidazole; Percutaneous drainage or aspiration of the liver abscess
  Arms: Cefixime plus Metronidazole Therapy

SUMMARY:
Liver abscess is purulent collections in the liver parenchyma that result from microbial infection spread to the liver through the biliary tree, hepatic or portal vein and by extension of adjacent infection or as a result of trauma. Liver abscesses are most commonly pyogenic followed by amoebic and rarely tuberculous or fungal in immunocompromised patients. In the developing country amoebic liver abscess is more frequent than the developed country but secondary bacterial infection of amoebic liver abscess and polymicrobial pyogenic liver abscess are also common.

Pyogenic liver abscess is commonly a polymicrobial infection caused by mixed enteric facultative and anaerobic pathogens. The most commonly isolated organisms are Escherichia coli, Klebsiella pneumoniae, Streptococcus constellatus, Streptococcus anginosus, Streptococcus intermedius, Enterococcus and anaerobes, including Bacteroidesfragilis and Fusobacteriumnecrophorum. Amoebic liver abscess most frequently occur following infection with the parasite Entamoeba histolytica.

Liver abscess is a common medical emergency. Prompt empirical antimicrobial with or without percutaneous aspiration or drainage of the abscess is therapeutic.

An empiric antimicrobial regimen for liver abscess should cover enteric gram-negative bacilli, streptococci, anaerobes and antamoebahistolytica. Presently a Fluoroquinolone (Ciprofloxacin, Levofloxacin) or a Third or Fourth generation Cefalosporine (Cefixime, Ceftriaxone, cefepime) or a Beta-lactam-beta-lactamase inhibitor combination (piperacillin-tazobactam or ticarcillin-clavulanate) or a Carbapenem (Imipenem-cilastatin, Meropenem, Doripenem, Ertapenem) are being used in combination with or without Metronidazole as the empirical antimicrobial regime for the treatment live abscess. There is no randomized controlled clinical trial to evaluated and compare efficacy of the antimicrobial regimens for the treatment of liver abscess as well as there is no specific treatment guideline for the use of empirical antibiotics. There is also no definite proven rational for using Cefalosporine, Beta-lactam-beta-lactamase inhibitor combination or Carbapenem upfront, not using Fluoroquinolone in empirical antibiotic regimen for the treatment of liver abscess. Injudicious use of broader spectrum antibiotics may also lead to rise in antibiotic resistance in future.

Both ciprofloxacin and Cefixime are effective oral antibiotics as they are well-absorbed orally with good oral bioavailability and achieve plasma concentration well above the minimal inhibitory concentrations require for the killing of the microorganism. Using intravenous (IV) antibiotics upfront, for the treatment of liver abscess in patients who can take orally may unnecessary increase the duration of hospital stay, healthcare burden and the cost of therapy, as well as the risk of hospital acquired infection.

So the investigators have planned this randomized controlled double blind study to evaluate the efficacy of empirical Ciprofloxacin plus Metronidazole and Cefixime plus Metronidazole therapy for the treatment of liver abscess and to compare the outcomes of two different empirical antibiotics regimen.

ELIGIBILITY:
Inclusion Criteria:

* Irrespective of gender
* Age ≥ 18 years
* Symptomatic patients of liver abscess confirmed with radiology imaging, either by ultrasonography (USG) or computed tomographgy (CT) scan

Exclusion Criteria:

* Past history of liver abscess
* Chronic kidney disease (CKD)
* History of hypersensitivity to either Ciprofloxacin or Metronidazole or Cefixime
* Shock (blood pressure <90/60 mmHg) at presentation
* ARDS (PaO2/FiO2≤300)
* Encephalopathy (altered sensorium with GCS <15)
* Acute kidney injury (AKI, Increase in serum creatinine to ≥1.5 times from the baseline)
* Pregnancy at presentation
* Already received antibiotics for more than 48 hours prior to the admission
* Not able to take orally
* Receiving blood thinners like anti-platelets, anti-coagulation agents within 4 weeks of presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Clinical cure | 2 weeks
  Asymptomatic and afebrile for more than 48 hours, along with USG showing no drainable collection in the liver with removal of the pigtail catheter if any

SECONDARY OUTCOMES:
Treatment failure | 8 weeks
  Defined as any one of the following condition
  1. Persistently symptomatic with fever for more than 72 hours even after starting empirical antibiotics and percutaneous aspiration or drainage
  2. Development of new collection in the liver during the course of antibiotic therapy
  3. Development of shock and new onset organ failure ( Encephalopathy, ARDS, AKI) during the course of therapy, leading to shifting to IV antibiotics
  4. If culture of the aspirated or drained pus show growth of microorganism not sensitive to either Ciprofloxacin or Cefixime
All-cause mortality | 8 weeks
  Total number of death
Recurrence of liver abscess | 8 weeks
  Development new liver abscess after clinical cure during the 8 weeks follow up period
Need for surgical intervention | 8 weeks
  number of patients needing surgical intervention for the treatment of liver abscess
Need for mechanical ventilation | 8 weeks
  Number of patients needing mechanical ventilation for the respiratory failure.
Need for prolong antibiotics 11. | 8 weeks
  Number of asymptomatic patients receiving 2 weeks of extended antibiotic therapy due to persistent drainage or aspiration even after 2 weeks of empirical antibiotics
Duration of hospital stay | 8 weeks
  Number of days of hospital stay for the treatment of liver abscess
Adverse drug events (ADE) | 8 weeks
  Number of adverse drug events
Localised bio-availability of the drugs (Ciprofloxacin, Metronidazole and Cefixime) | 8 weeks
  Concentration of the drug in drained pus/Concentration of drug in the serum X100 on the day-three of the drainage (when applicable)

CONTACTS AND LOCATIONS:
Overall Officials: Deba P Dhibar, MD, Principal Investigator — PGIMER, Chandigarh, India
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers except for those are directly involved with this study.

REFERENCES:
- [Derived] Priya G L, Dhibar DP, Saroch A, Sharma N, Sharma V, Verma N, Chaluvashetty SB, Prakash A, Kaur H. Efficacy of empirical Ciprofloxacin or Cefixime plus Metronidazole therapy for the treatment of liver abscess: a randomized control clinical trial. Sci Rep. 2024 May 20;14(1):11430. doi: 10.1038/s41598-024-59607-1. PMID 38769330